CLINICAL TRIAL: NCT03308968
Title: A Multicenter, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Study With an Open-Label Period to Evaluate the Efficacy and Safety of Fremanezumab for the Prophylactic Treatment of Migraine in Patients With Inadequate Response to Prior Preventive Treatments
Brief Title: An Efficacy and Safety Study of Fremanezumab in Adults With Migraine
Acronym: FOCUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TV48125-CNS-30068; 2017-002441-30 (EudraCT Number)
Expanded Access: NCT03539393 (Available)
Record Dates: First submitted 2017-10-03; First posted 2017-10-13 (Actual); Results first posted 2019-10-09 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Migraine Prophylaxis
MeSH Terms: interventions — fremanezumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Double-blind (DB) period: Participants with CM or EM will receive 3 injections of placebo 1.5 milliliters (mL) SC on Day 0 and single injection of placebo 1.5 mL SC on Days 28 and 56. Open-label (OL) period: Participants with CM or EM will receive fremanezumab (TEV-48125) 225 milligrams (mg) SC (1 injection of fremanezumab 225 mg/1.5 mL) at Days 84, 112, and 140.
  Interventions: Drug: Fremanezumab; Drug: Placebo
- Fremanezumab Quarterly (Experimental): DB period: Participants with CM or EM will receive fremanezumab 675 mg SC (3 injections of fremanezumab 225 mg/1.5 mL) on Day 0 followed by monthly SC administration of placebo 1.5 mL for 2 months (on Days 28 and 56). OL period: Participants with CM or EM will receive fremanezumab 225 mg SC (1 injection of fremanezumab 225 mg/1.5 mL) at Days 84, 112, and 140.
  Interventions: Drug: Fremanezumab; Drug: Placebo
- Fremanezumab Monthly (Experimental): DB period: Participants with CM will receive fremanezumab 675 mg SC (3 injections of fremanezumab 225 mg/1.5 mL) on Day 0 followed by monthly SC administration of fremanezumab 225 mg (1 injection of fremanezumab 225 mg/1.5 mL) for 2 months (on Days 28 and 56). Participants with EM will receive fremanezumab 225 mg SC (1 injection of fremanezumab 225 mg/1.5 mL and 2 injections of placebo 1.5 mL) on Day 0 followed by monthly SC administration of fremanezumab 225 mg (1 injection of fremanezumab 225 mg/1.5 mL) for 2 months (on Days 28 and 56). OL period: Participants with CM or EM will receive fremanezumab 225 mg SC (1 injection of fremanezumab 225 mg/1.5 mL) at Days 84, 112, and 140.
  Interventions: Drug: Fremanezumab; Drug: Placebo

INTERVENTIONS:
Drug: Fremanezumab — Fremanezumab will be administered per dose and schedule specified in the arm.
  Other Names: TEV-48125
Drug: Placebo — Placebo matching to fremanezumab will be administered per schedule specified in the arm.

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and tolerability of monthly and quarterly subcutaneous (sc) injections of fremanezumab compared with sc injections of placebo in participants with chronic migraine (CM) or episodic migraine (EM) who have responded inadequately to 2 to 4 classes of prior preventive treatments.

Approximately equal numbers of participants from each subgroup (CM and EM) are randomized in blinded-fashion 1:1:1 into one of 3 treatments for the subgroup - 2 active treatments and 1 placebo treatment- consisting of monthly injections for 3 months (up to Week 12). Then all participants continue into an open-label extension of 3 months (up to Week 24) during which everyone is administered sc injections of fremanezumab.

ELIGIBILITY:
Inclusion Criteria:

* The participant has a diagnosis of migraine with onset at ≤50 years of age.
* Body weight ≥45 kilograms.
* The participant has a history of migraine for ≥12 months prior to screening.
* Women of childbearing potential (WOCBP) whose male partners are potentially fertile (that is; no vasectomy) must use highly effective birth control methods for the duration of the study and the follow-up period and for 6.0 months after discontinuation of investigational medicinal product (IMP)
* Men must be sterile, or if they are potentially fertile/reproductively competent (not surgically [that is; vasectomy] or congenitally sterile) and their female partners are of childbearing potential, must use, together with their female partners, acceptable birth control methods for the duration of the study and for 6.0 months after discontinuation of the investigational medicinal product (IMP).

  * Additional criteria apply, please contact the investigator for more information.

Exclusion Criteria:

* At the time of screening visit, participant is receiving any preventive migraine medications, regardless of the medical indication for more than 5 days and expects to continue with these medications.
* Participant has received onabotulinumtoxinA for migraine or for any medical or cosmetic reasons requiring injections in the head, face, or neck during the 3 months before screening visit.
* The participant has used an intervention/device (for example; scheduled nerve blocks and transcranial magnetic stimulation) for migraine during the 2 months prior to screening.
* The participant uses triptans/ergots as preventive therapies for migraine.
* Participant uses non-steroidal anti-inflammatory drugs (NSAIDs) as preventive therapy for migraine on nearly daily basis for other indications. Note: Low dose aspirin (for example; 81 mg) used for cardiovascular disease prevention is allowed.

  * Additional criteria apply, please contact the investigator for more information.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 838 (Actual)
Dates: Start 2017-10-13 (Actual); Primary Completion 2018-10-02 (Actual); Study Completion 2019-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (113):
- United States (30):
  - Teva Investigational Site 14742, Huntsville, Alabama
  - Teva Investigational Site 14729, Long Beach, California
  - Teva Investigational Site 14739, San Diego, California
  - Teva Investigational Site 14843, Santa Monica, California
  - Teva Investigational Site 14749, Colorado Springs, Colorado
  - Teva Investigational Site 14758, Maitland, Florida
  - Teva Investigational Site 14738, Orlando, Florida
  - Teva Investigational Site 14760, Decatur, Georgia
  - Teva Investigational Site 14737, Meridian, Idaho
  - Teva Investigational Site 14730, Chicago, Illinois
  - Teva Investigational Site 14740, Evanston, Illinois
  - Teva Investigational Site 14735, Louisville, Kentucky
  - Teva Investigational Site 14747, Pikesville, Maryland
  - Teva Investigational Site 14750, Fall River, Massachusetts
  - Teva Investigational Site 14734, Watertown, Massachusetts
  - Teva Investigational Site 14731, Ann Arbor, Michigan
  - Teva Investigational Site 14748, Plymouth, Minnesota
  - Teva Investigational Site 14746, Omaha, Nebraska
  - Teva Investigational Site 14754, Berlin, New Jersey
  - Teva Investigational Site 14752, Albuquerque, New Mexico
  - Teva Investigational Site 14753, Amherst, New York
  - Teva Investigational Site 14736, Greensboro, North Carolina
  - Teva Investigational Site 14741, Greensboro, North Carolina
  - Teva Investigational Site 14732, Raleigh, North Carolina
  - Teva Investigational Site 14761, Lincoln, Rhode Island
  - Teva Investigational Site 14756, Warwick, Rhode Island
  - Teva Investigational Site 14745, Memphis, Tennessee
  - Teva Investigational Site 14743, Nashville, Tennessee
  - Teva Investigational Site 14733, Austin, Texas
  - Teva Investigational Site 14751, West Jordan, Utah
- Belgium (4):
  - Teva Investigational Site 37092, Bruges
  - Teva Investigational Site 37089, Brussels
  - Teva Investigational Site 37091, Hasselt
  - Teva Investigational Site 37090, Liège
- Czechia (10):
  - Teva Investigational Site 54162, Brno
  - Teva Investigational Site 54159, Ostrava
  - Teva Investigational Site 54165, Ostrava-Moravska
  - Teva Investigational Site 54158, Pardubice
  - Teva Investigational Site 54163, Prague
  - Teva Investigational Site 54161, Prague
  - Teva Investigational Site 54164, Prague
  - Teva Investigational Site 54160, Prague
  - Teva Investigational Site 54166, Prague
  - Teva Investigational Site 54157, Rychnov nad Kněžnou
- Denmark (5):
  - Teva Investigational Site 39051, Aalborg
  - Teva Investigational Site 39049, Aarhus
  - Teva Investigational Site 39052, Ballerup Municipality
  - Teva Investigational Site 39048, Glostrup Municipality
  - Teva Investigational Site 39050, Vejle
- Finland (6):
  - Teva Investigational Site 40034, Helsinki
  - Teva Investigational Site 40035, Helsinki
  - Teva Investigational Site 40036, Oulu
  - Teva Investigational Site 40033, Tampere
  - Teva Investigational Site 40032, Turku
  - Teva Investigational Site 40037, Turku
- France (6):
  - Teva Investigational Site 35237, Bron
  - Teva Investigational Site 35238, Lille
  - Teva Investigational Site 35235, Marseille
  - Teva Investigational Site 35240, Nice
  - Teva Investigational Site 35239, Strasbourg
  - Teva Investigational Site 35236, Voiron
- Germany (12):
  - Teva Investigational Site 32697, Berlin
  - Teva Investigational Site 32690, Berlin
  - Teva Investigational Site 32694, Bochum
  - Teva Investigational Site 32699, Essen
  - Teva Investigational Site 32692, Göppingen
  - Teva Investigational Site 32691, Halle
  - Teva Investigational Site 32698, Hamburg
  - Teva Investigational Site 32700, Kiel
  - Teva Investigational Site 32695, Königstein im Taunus
  - Teva Investigational Site 32689, München
  - Teva Investigational Site 32701, Rostock
  - Teva Investigational Site 32693, Ulm
- Italy (2):
  - Teva Investigational Site 30199, Florence
  - Teva Investigational Site 30204, Roma
- Netherlands (4):
  - Teva Investigational Site 38126, Amsterdam
  - Teva Investigational Site 38127, Blaricum
  - Teva Investigational Site 38124, Leiden
  - Teva Investigational Site 38125, Tilburg
- Poland (9):
  - Teva Investigational Site 53420, Krakow
  - Teva Investigational Site 53425, Krakow
  - Teva Investigational Site 53422, Lodz
  - Teva Investigational Site 53424, Lodz
  - Teva Investigational Site 53418, Lublin
  - Teva Investigational Site 53416, Poznan
  - Teva Investigational Site 53419, Szczecin
  - Teva Investigational Site 53417, Warsaw
  - Teva Investigational Site 53423, Warsaw
- Spain (11):
  - Teva Investigational Site 31231, Barcelona
  - Teva Investigational Site 31235, Madrid
  - Teva Investigational Site 31236, Madrid
  - Teva Investigational Site 31226, Pamplona
  - Teva Investigational Site 31229, Santander
  - Teva Investigational Site 31230, Santiago de Compostela
  - Teva Investigational Site 31234, Seville
  - Teva Investigational Site 31233, Valencia
  - Teva Investigational Site 31227, Valencia
  - Teva Investigational Site 31225, Valladolid
  - Teva Investigational Site 31228, Zaragoza
- Sweden (5):
  - Teva Investigational Site 42050, Helsingborg
  - Teva Investigational Site 42049, Huddinge
  - Teva Investigational Site 42051, Lund
  - Teva Investigational Site 42052, Stockholm
  - Teva Investigational Site 42054, Stockholm
- Switzerland (3):
  - Teva Investigational Site 45018, Bad Zurzach
  - Teva Investigational Site 45016, Bern
  - Teva Investigational Site 45017, Lugano
- United Kingdom (6):
  - Teva Investigational Site 34231, Glasgow
  - Teva Investigational Site 34232, Hull
  - Teva Investigational Site 34233, London
  - Teva Investigational Site 34230, Oxford
  - Teva Investigational Site 34235, Salford
  - Teva Investigational Site 34236, Stoke-on-Trent

REFERENCES:
- [Derived] McAllister P, Cohen JM, Campos VR, Ning X, Janka L, Barash S. Impact of fremanezumab on disability outcomes in patients with episodic and chronic migraine: a pooled analysis of phase 3 studies. J Headache Pain. 2022 Aug 29;23(1):112. doi: 10.1186/s10194-022-01438-4. PMID 36038833
- [Derived] Diener HC, McAllister P, Jurgens TP, Kessler Y, Ning X, Cohen JM, Campos VR, Barash S, Silberstein SD. Safety and tolerability of fremanezumab in patients with episodic and chronic migraine: a pooled analysis of phase 3 studies. Cephalalgia. 2022 Jul;42(8):769-780. doi: 10.1177/03331024221076485. Epub 2022 Mar 25. PMID 35331009
- [Derived] Lampl C, Rapoport AM, Cohen JM, Barash S, Ramirez Campos V, Seminerio MJ, Ning X, Silberstein SD. Efficacy and quality-of-life improvements with fremanezumab treatment in patients with difficult-to-treat migraine with associated neurological dysfunction. Eur J Neurol. 2022 Jul;29(7):2129-2137. doi: 10.1111/ene.15328. Epub 2022 Mar 29. PMID 35302681
- [Derived] MaassenVanDenBrink A, Terwindt GM, Cohen JM, Barash S, Campos VR, Galic M, Ning X, Karppa M. Impact of age and sex on the efficacy of fremanezumab in patients with difficult-to-treat migraine: results of the randomized, placebo-controlled, phase 3b FOCUS study. J Headache Pain. 2021 Dec 18;22(1):152. doi: 10.1186/s10194-021-01336-1. PMID 34922436
- [Derived] Nahas SJ, Naegel S, Cohen JM, Ning X, Janka L, Campos VR, Krasenbaum LJ, Holle-Lee D, Kudrow D, Lampl C. Efficacy and safety of fremanezumab in clinical trial participants aged >/=60 years with episodic or chronic migraine: pooled results from 3 randomized, double-blind, placebo-controlled phase 3 studies. J Headache Pain. 2021 Nov 24;22(1):141. doi: 10.1186/s10194-021-01351-2. PMID 34819017
- [Derived] Ashina M, Cohen JM, Galic M, Campos VR, Barash S, Ning X, Kessler Y, Janka L, Diener HC. Efficacy and safety of fremanezumab in patients with episodic and chronic migraine with documented inadequate response to 2 to 4 classes of migraine preventive medications over 6 months of treatment in the phase 3b FOCUS study. J Headache Pain. 2021 Jul 10;22(1):68. doi: 10.1186/s10194-021-01279-7. PMID 34246226
- [Derived] Pazdera L, Cohen JM, Ning X, Campos VR, Yang R, Pozo-Rosich P. Fremanezumab for the Preventive Treatment of Migraine: Subgroup Analysis by Number of Prior Preventive Treatments with Inadequate Response. Cephalalgia. 2021 Sep;41(10):1075-1088. doi: 10.1177/03331024211008401. Epub 2021 May 14. PMID 33990144
- [Derived] Spierings ELH, Karppa M, Ning X, Cohen JM, Campos VR, Yang R, Reuter U. Efficacy and safety of fremanezumab in patients with migraine and inadequate response to prior preventive treatment: subgroup analyses by country of a randomized, placebo-controlled trial. J Headache Pain. 2021 Apr 16;22(1):26. doi: 10.1186/s10194-021-01232-8. PMID 33863272
- [Derived] Ferrari MD, Diener HC, Ning X, Galic M, Cohen JM, Yang R, Mueller M, Ahn AH, Schwartz YC, Grozinski-Wolff M, Janka L, Ashina M. Fremanezumab versus placebo for migraine prevention in patients with documented failure to up to four migraine preventive medication classes (FOCUS): a randomised, double-blind, placebo-controlled, phase 3b trial. Lancet. 2019 Sep 21;394(10203):1030-1040. doi: 10.1016/S0140-6736(19)31946-4. Epub 2019 Aug 16. PMID 31427046

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 838 participants were randomized in a 1:1:1 ratio to placebo, fremanezumab quarterly, or fremanezumab monthly treatment groups.
Groups:
- Placebo: Double-blind (DB) period: Participants with chronic migraine (CM) or episodic migraine (EM) received 3 injections of placebo 1.5 milliliters (mL) subcutaneously (SC) on Day 0 and single injection of placebo 1.5 mL SC on Days 28 and 56. Open-label (OL) period: Participants with CM or EM received fremanezumab (TEV-48125) 225 milligrams (mg) SC (1 injection of fremanezumab 225 mg/1.5 mL) at Days 84, 112, and 140.
- Fremanezumab Quarterly: DB period: Participants with CM or EM received fremanezumab 675 mg SC (3 injections of fremanezumab 225 mg/1.5 mL) on Day 0 followed by monthly SC administration of placebo 1.5 mL for 2 months (on Days 28 and 56). OL period: Participants with CM or EM received fremanezumab 225 mg SC (1 injection of fremanezumab 225 mg/1.5 mL) at Days 84, 112, and 140.
- Fremanezumab Monthly: DB period: Participants with CM received fremanezumab 675 mg SC (3 injections of fremanezumab 225 mg/1.5 mL) on Day 0 followed by monthly SC administration of fremanezumab 225 mg (1 injection of fremanezumab 225 mg/1.5 mL) for 2 months (on Days 28 and 56). Participants with EM received fremanezumab 225 mg SC (1 injection of fremanezumab 225 mg/1.5 mL and 2 injections of placebo 1.5 mL) on Day 0 followed by monthly SC administration of fremanezumab 225 mg (1 injection of fremanezumab 225 mg/1.5 mL) for 2 months (on Days 28 and 56).OL period: Participants with CM or EM received fremanezumab 225 mg SC (1 injection of fremanezumab 225 mg/1.5 mL) at Days 84, 112, and 140.
Period: Double-Blind Period (12 Weeks)
Arm/Group | Placebo | Fremanezumab Quarterly | Fremanezumab Monthly
Started (Intent-to-treat (ITT) analysis set: all randomized participants.) | 279 | 276 | 283
DB Safety Analysis Set (Participants who received at least 1 dose of study drug during DB period.) | 277 (2 participants (1 with CM and 1 with EM) randomized to placebo but received Fremanezumab monthly.) | 276 | 285 (2 participants (1 with CM and 1 with EM) randomized to placebo but received Fremanezumab monthly.)
DB Modified ITT (mITT) Analysis Set (Received ≥1 dose of study drug;had ≥10 days of postbaseline efficacy assessment on primary endpoint.) | 278 | 276 | 283
Completed | 264 | 271 | 272
Not Completed | 15 | 5 | 11
Not completed — Adverse Event | 3 | 1 | 4
Not completed — Withdrawal by Subject | 2 | 2 | 3
Not completed — Protocol Violation | 6 | 0 | 2
Not completed — Non-compliance to study procedures | 1 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 1 | 0
Not completed — Other than specified | 1 | 0 | 2
Period: Open-Label Period (12 Weeks)
Arm/Group | Placebo | Fremanezumab Quarterly | Fremanezumab Monthly
Started (OL Safety analysis set: Participants who received at least 1 dose of study drug during OL period.) | 264 | 271 | 272
OL mITT Analysis Set (Received ≥1 dose of study drug in OL period;had ≥10 days of postbaseline diary entries in OL period.) | 263 | 271 | 272
Completed | 253 | 259 | 260
Not Completed | 11 | 12 | 12
Not completed — Other than specified | 1 | 2 | 1
Not completed — Adverse Event | 4 | 1 | 1
Not completed — Withdrawal by Subject | 5 | 5 | 7
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Non-compliance to study procedures | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Lack of Efficacy | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Population: ITT analysis set included all randomized participants.
Groups:
- Placebo: DB period: Participants with CM or EM received 3 injections of placebo 1.5 mL SC on Day 0 and single injection of placebo 1.5 mL SC on Days 28 and 56. OL period: Participants with CM or EM received fremanezumab (TEV-48125) 225 mg SC (1 injection of fremanezumab 225 mg/1.5 mL) at Days 84, 112, and 140.
- Fremanezumab Monthly: DB period: Participants with CM received fremanezumab 675 mg SC (3 injections of fremanezumab 225 mg/1.5 mL) on Day 0 followed by monthly SC administration of fremanezumab 225 mg (1 injection of fremanezumab 225 mg/1.5 mL) for 2 months (on Days 28 and 56). Participants with EM received fremanezumab 225 mg SC (1 injection of fremanezumab 225 mg/1.5 mL and 2 injections of placebo 1.5 mL) on Day 0 followed by monthly SC administration of fremanezumab 225 mg (1 injection of fremanezumab 225 mg/1.5 mL) for 2 months (on Days 28 and 56). OL period: Participants with CM or EM received fremanezumab 225 mg SC (1 injection of fremanezumab 225 mg/1.5 mL) at Days 84, 112, and 140.
- Total: Total of all reporting groups
Arm/Group | Placebo | Fremanezumab Quarterly | Fremanezumab Monthly | Total
Number analyzed (Participants) | 279 | 276 | 283 | 838
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.8 (11.10) | 45.8 (10.97) | 45.9 (11.05) | 46.2 (11.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 233 | 229 | 238 | 700
  Male | 46 | 47 | 45 | 138
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 6 | 7 | 24
  Not Hispanic or Latino | 255 | 260 | 264 | 779
  Unknown or Not Reported | 13 | 10 | 12 | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 1 | 0 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 4 | 8
  White | 262 | 262 | 262 | 786
  Other | 1 | 2 | 1 | 4
  Unknown or Not Reported | 13 | 10 | 12 | 35
Number of Migraine Days During the 28 Day Baseline Period [Mean (Standard Deviation); unit: days] — A migraine day was defined as when at least 1 of the following situations occurred: A calendar day (0:00 to 23:59) demonstrating at least 4 consecutive hours of a headache meeting criteria for migraine with or without aura; a calendar day (0:00 to 23:59) demonstrating at least 4 consecutive hours of a headache meeting criteria for probable migraine, a migraine subtype where only 1 migraine criterion was missing; a calendar day (0:00 to 23:59) demonstrating a headache of any duration that was treated with migraine-specific medications (triptans and ergot compounds). Population: Here, 'Number analyzed' signifies participants evaluable for this measure.
  days
    number analyzed (Participants) | 279 | 275 | 283 | 837
    (all) | 14.3 (6.12) | 14.1 (5.61) | 14.1 (5.58) | 14.2 (5.77)
Number of Headache Days of at Least Moderate Severity During the 28 Day Baseline Period [Mean (Standard Deviation); unit: days] — Headaches were subjectively rated by participants as mild, moderate or severe. A headache day of at least moderate severity was defined as a calendar day (00:00 to 23:59) demonstrating at least 4 consecutive hours of headache of at least moderate severity or; a calendar day (0:00 to 23:59) demonstrating a headache of any duration that was treated with migraine-specific acute medications (triptans and ergot compounds). Population: Here, 'Number analyzed' signifies participants evaluable for this measure.
  days
    number analyzed (Participants) | 279 | 275 | 283 | 837
    (all) | 12.8 (5.92) | 12.4 (5.84) | 12.7 (5.82) | 12.6 (5.85)

OUTCOME MEASURES:

1. Primary Outcome: DB Period: Change From Baseline in Monthly Average Number of Migraine Days During the 12-Week Period After the First Dose of Fremanezumab
Description: A migraine day was defined as when at least 1 of the following situations occurred: A calendar day (0:00 to 23:59) demonstrating at least 4 consecutive hours of a headache meeting criteria for migraine with or without aura; a calendar day (0:00 to 23:59) demonstrating at least 4 consecutive hours of a headache meeting criteria for probable migraine, a migraine subtype where only 1 migraine criterion was missing; a calendar day (0:00 to 23:59) demonstrating a headache of any duration that was treated with migraine-specific medications (triptans and ergot compounds). Monthly averages were derived and normalized to 28 days equivalent by formula: (number of days of efficacy variable over relevant period/number of days with assessments recorded in e-diary over relevant period)*28. Change was calculated as post-baseline value - baseline value.
Time Frame: Baseline (Day -28 to Day -1), up to Week 12
Population: DB mITT analysis set included participants who received at least 1 dose of study drug and had at least 10 days of postbaseline efficacy assessment on the primary endpoint.
Measure: Least Squares Mean (Standard Error); unit: days/month
Groups:
- Placebo: DB period: Participants with CM or EM received 3 injections of placebo 1.5 mL SC on Day 0 and single injection of placebo 1.5 mL SC on Days 28 and 56.
- Fremanezumab Quarterly: DB period: Participants with CM or EM received fremanezumab 675 mg SC (3 injections of fremanezumab 225 mg/1.5 mL) on Day 0 followed by monthly SC administration of placebo 1.5 mL for 2 months (on Days 28 and 56).
- Fremanezumab Monthly: DB period: Participants with CM received fremanezumab 675 mg SC (3 injections of fremanezumab 225 mg/1.5 mL) on Day 0 followed by monthly SC administration of fremanezumab 225 mg (1 injection of fremanezumab 225 mg/1.5 mL) for 2 months (on Days 28 and 56). Participants with EM received fremanezumab 225 mg SC (1 injection of fremanezumab 225 mg/1.5 mL and 2 injections of placebo 1.5 mL) on Day 0 followed by monthly SC administration of fremanezumab 225 mg (1 injection of fremanezumab 225 mg/1.5 mL) for 2 months (on Days 28 and 56).
Arm/Group | Placebo | Fremanezumab Quarterly | Fremanezumab Monthly
Number analyzed (Participants) | 278 | 276 | 283
days/month | -0.6 (0.34) | -3.7 (0.34) | -4.1 (0.34)
Statistical Analysis 1: Comparison: Placebo vs Fremanezumab Quarterly; Analysis was performed using analysis of covariance (ANCOVA) method with treatment, sex, region, special group of treatment failure (yes or no), migraine classification (that is; CM or EM), and treatment-by-migraine classification interaction as fixed effects, and baseline number of migraine days and years since onset of migraines as covariates. The stratification factors (as randomized) were used in the model; Test type: Other; p < 0.0001, ANCOVA; Least square (LS) mean difference = -3.1, 95% CI 2-sided [-3.84 to -2.42], Standard Error of Mean 0.36
Statistical Analysis 2: Comparison: Placebo vs Fremanezumab Monthly; Analysis was performed using ANCOVA method with treatment, sex, region, special group of treatment failure (yes or no), migraine classification (that is; CM or EM), and treatment-by-migraine classification interaction as fixed effects, and baseline number of migraine days and years since onset of migraines as covariates. The stratification factors (as randomized) were used in the model; Test type: Other; p < 0.0001, ANCOVA; LS mean difference = -3.5, 95% CI 2-sided [-4.19 to -2.78], Standard Error of Mean 0.36

2. Secondary Outcome: DB Period: Percentage of Participants Reaching at Least 50 Percent (%) Reduction From Baseline in Monthly Average Number of Migraine Days During the 12-Week Period After the First Dose of Fremanezumab
Description: A migraine day was defined as when at least 1 of the following situations occurred: A calendar day (0:00 to 23:59) demonstrating at least 4 consecutive hours of a headache meeting criteria for migraine with or without aura; a calendar day (0:00 to 23:59) demonstrating at least 4 consecutive hours of a headache meeting criteria for probable migraine, a migraine subtype where only 1 migraine criterion was missing; a calendar day (0:00 to 23:59) demonstrating a headache of any duration that was treated with migraine-specific medications (triptans and ergot compounds). Monthly averages were derived and normalized to 28 days equivalent by formula: (number of days of efficacy variable over relevant period/number of days with assessments recorded in e-diary over relevant period)*28.
Time Frame: Baseline (Day -28 to Day-1), up to Week 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Fremanezumab Quarterly | Fremanezumab Monthly
Number analyzed (Participants) | 278 | 276 | 283
percentage of participants | 9 | 34 | 34

3. Secondary Outcome: DB Period: Change From Baseline in Monthly Average Number of Headache Days of at Least Moderate Severity During the 12-Week Period After the First Dose of Fremanezumab
Description: A headache day of at least moderate severity was defined as a calendar day (00:00 to 23:59) demonstrating at least 4 consecutive hours of headache of at least moderate severity or; a calendar day (0:00 to 23:59) demonstrating a headache of any duration that was treated with migraine-specific acute medications (triptans and ergot compounds). Monthly averages were derived and normalized to 28 days equivalent by the following formula: (number of days of efficacy variable over relevant period/number of days with assessments recorded in the e-diary over the relevant period) * 28. The change was calculated as post-baseline value - baseline value. LS mean calculated using ANCOVA model with treatment, gender, region, special group of treatment failure (yes/no), migraine classification (EM/CM), and treatment*migraine classification as fixed effects and baseline number of headache days of at least moderate severity and years since onset of migraine as covariates.
Time Frame: Baseline (Day -28 to Day -1), up to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: days/month
Arm/Group | Placebo | Fremanezumab Quarterly | Fremanezumab Monthly
Number analyzed (Participants) | 278 | 276 | 283
days/month | -0.6 (0.33) | -3.9 (0.34) | -4.2 (0.34)

4. Secondary Outcome: DB Period: Change From Baseline in Monthly Average Number of Migraine Days During the 4-Week Period After the First Dose of Fremanezumab
Description: A migraine day was defined as when at least 1 of following occurred: A calendar day (0:00 to 23:59) demonstrating at least 4 consecutive hours of a headache meeting criteria for migraine with or without aura; a calendar day demonstrating at least 4 consecutive hours of a headache meeting criteria for probable migraine, a migraine subtype where only 1 migraine criterion was missing; a calendar day demonstrating a headache of any duration that was treated with migraine-specific medications. Monthly averages were derived and normalized to 28 days equivalent by formula: (number of days of efficacy variable over relevant period/number of days with assessments recorded in e-diary over relevant period)*28. LS mean calculated using ANCOVA model with treatment, gender, region, special group of treatment failure (yes/no), migraine classification (EM/CM), and treatment*migraine classification as fixed effects, and baseline number of migraine days and years since onset of migraines as covariates.
Time Frame: Baseline (Day -28 to Day -1), up to Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: days/month
Arm/Group | Placebo | Fremanezumab Quarterly | Fremanezumab Monthly
Number analyzed (Participants) | 278 | 276 | 283
days/month | -0.6 (0.35) | -4.1 (0.35) | -4.1 (0.35)

5. Secondary Outcome: DB Period: Percentage of Participants Reaching at Least 50% Reduction From Baseline in Monthly Average Number of Migraine Days During the 4-Week Period After the First Dose of Fremanezumab
Description: as for outcome 2
Time Frame: Baseline (Day -28 to Day-1), up to Week 4
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Fremanezumab Quarterly | Fremanezumab Monthly
Number analyzed (Participants) | 278 | 276 | 283
percentage of participants | 10 | 38 | 36

6. Secondary Outcome: DB Period: Change From Baseline in Monthly Average Number of Days of Use of Any Acute Headache Medications During the 12-Week Period After the First Dose of Fremanezumab
Description: Baseline data and the mean change from baseline in the monthly average number of days of use of any acute headache medications during the 12-week period after administration of the first dose of study drug (based on Week 0 to 12 data) is reported. Least Squares (LS) mean calculated using analysis of covariance (ANCOVA) model with treatment, gender, region, special group of treatment failure (yes/no), migraine classification (EM/CM), and treatment*migraine classification as fixed effects, and baseline number of migraine days and years since onset of migraines as covariates.
Time Frame: Baseline (Day -28 to Day -1), up to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: days/month
Arm/Group | Placebo | Fremanezumab Quarterly | Fremanezumab Monthly
Number analyzed (Participants) | 278 | 276 | 283
days/month | -0.6 (0.32) | -3.7 (0.32) | -3.9 (0.32)

7. Secondary Outcome: DB Period: Change From Baseline in Monthly Average Number of Headache Days of at Least Moderate Severity During the 4-Week Period After the First Dose of Fremanezumab
Description: A headache day of at least moderate severity was defined as a calendar day (00:00 to 23:59) demonstrating at least 4 consecutive hours of headache of at least moderate severity or; a calendar day (0:00 to 23:59) demonstrating a headache of any duration that was treated with migraine-specific acute medications (triptans and ergot compounds). Monthly averages were derived and normalized to 28 days equivalent by the following formula: (number of days of efficacy variable over relevant period/number of days with assessments recorded in the e-diary over the relevant period) * 28. The change was calculated as post-baseline value - baseline value. LS mean calculated using ANCOVA model with treatment, gender, region, special group of treatment failure (yes/no), migraine classification (EM/CM), and treatment*migraine classification as fixed effects, and baseline number of headache days of at least moderate severity and years since onset of migraines as covariates.
Time Frame: Baseline (Day -28 to Day -1), up to Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: days/month
Arm/Group | Placebo | Fremanezumab Quarterly | Fremanezumab Monthly
Number analyzed (Participants) | 278 | 276 | 283
days/month | -0.5 (0.34) | -4.2 (0.35) | -4.5 (0.34)

8. Secondary Outcome: DB Period: Number of Participants With Adverse Events (AEs) and Who Did Not Complete the Study Due to AEs
Description: An AE was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Severe AE was defined as inability to carry out usual activities. Treatment-related AEs were defined as AEs with possible, probable, definite, or missing relationship to study drug. Serious AEs were defined as death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized participant and required medical intervention to prevent 1 of the outcomes listed in this definition. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline (Day 0) up to Week 12
Population: DB safety analysis set included all randomized participants who received at least 1 dose of study drug during the DB treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab Quarterly | Fremanezumab Monthly
Number analyzed (Participants) | 277 | 276 | 285
Participants
  Any AEs | 134 | 151 | 129
  AEs leading to withdrawal from study | 3 | 1 | 4

9. Secondary Outcome: OL Period: Number of Participants With AEs and Who Did Not Complete the Study Due to AEs
Description: as for outcome 8
Time Frame: Week 12 up to Week 24
Population: OL safety analysis set included all participants who received at least 1 dose of study drug during the OL treatment period.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo; Fremanezumab Quarterly; Fremanezumab Monthly: OL period: Participants with CM or EM received fremanezumab 225 mg SC (1 injection of fremanezumab 225 mg/1.5 mL) at Days 84, 112, and 140.
Arm/Group | Placebo | Fremanezumab Quarterly | Fremanezumab Monthly
Number analyzed (Participants) | 262 | 271 | 274
Participants
  Any AEs | 137 | 149 | 155
  AEs leading to withdrawal from study | 4 | 1 | 2

10. Secondary Outcome: DB Period: Number of Participants With Potentially Clinically Significant Abnormal Serum Chemistry Results
Description: Criteria for potentially clinically significant abnormal serum chemistry values included: alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), gamma glutamyl transferase (GGT), and lactate dehydrogenase (LDH) (units/liter [U/L]): greater than or equal to (≥) 3*upper limit of normal (ULN); Blood Urea Nitrogen (BUN): ≥10.71 millimoles/liter (mmol/L); creatinine: ≥177 micromoles/liter (µmol/L); bilirubin (total): ≥34.2 µmol/L; and uric acid: ≥625 µmol/L (men), and ≥506 µmol/L (women). A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline up to Week 12
Population: DB safety analysis set included all randomized participants who received at least 1 dose of study drug during the DB treatment period. Here, 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab Quarterly | Fremanezumab Monthly
Number analyzed (Participants) | 272 | 268 | 280
Participants | 1 | 3 | 4

11. Secondary Outcome: OL Period: Number of Participants With Potentially Clinically Significant Abnormal Serum Chemistry Results
Description: Criteria for potentially clinically significant abnormal serum chemistry values included: ALT, AST, ALP, GGT, and LDH (U/L): ≥3*ULN; BUN: ≥10.71 mmol/L; creatinine: ≥177 µmol/L; bilirubin (total): ≥34.2 µmol/L; and uric acid: ≥625 µmol/L (men), and ≥506 µmol/L (women). A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Week 12 up to Week 24
Population: OL safety analysis set included all participants who received at least 1 dose of study drug during the OL treatment period. Here, 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab Quarterly | Fremanezumab Monthly
Number analyzed (Participants) | 259 | 270 | 273
Participants | 2 | 3 | 2

12. Secondary Outcome: DB Period: Number of Participants With Potentially Clinically Significant Abnormal Hematology Results
Description: Criteria for potentially clinically significant abnormal hematology values included: hemoglobin: less than (<) 115 grams/liter (g/L) (in men) or less than or equal to (≤) 95 g/L (in women), hematocrit: <0.37 L/L (in men) or <0.32 L/L (in women), leukocytes: ≥20*10^9/L or ≤3*10^9/L, eosinophils: >=10%, platelets: ≥700*10^9/L or ≤75*10^9/L, and absolute neutrophil count (ANC): ≤1*10^9/L. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline up to Week 12
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab Quarterly | Fremanezumab Monthly
Number analyzed (Participants) | 271 | 268 | 278
Participants | 11 | 12 | 3

13. Secondary Outcome: OL Period: Number of Participants With Potentially Clinically Significant Abnormal Hematology Results
Description: Criteria for potentially clinically significant abnormal hematology values included: hemoglobin: <115 g/L (in men) or ≤95 g/L (in women), hematocrit: <0.37 L/L (in men) or <0.32 L/L (in women), leukocytes: ≥20*10^9/L or ≤3*10^9/L, eosinophils: >=10%, platelets: ≥700*10^9/L or ≤75*10^9/L, and ANC: ≤1*10^9/L. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Week 12 up to Week 24
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab Quarterly | Fremanezumab Monthly
Number analyzed (Participants) | 259 | 270 | 273
Participants | 9 | 11 | 5

14. Secondary Outcome: DB Period: Number of Participants With Potentially Clinically Significant Abnormal Coagulation Laboratory Test Results
Description: Criteria for potentially clinically significant abnormal coagulation values included: prothrombin international normalized ratio (INR): greater than (>) 1.5. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline up to Week 12
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab Quarterly | Fremanezumab Monthly
Number analyzed (Participants) | 269 | 267 | 277
Participants | 2 | 4 | 4

15. Secondary Outcome: OL Period: Number of Participants With Potentially Clinically Significant Abnormal Coagulation Laboratory Test Results
Description: Criteria for potentially clinically significant abnormal coagulation values included: prothrombin INR: >1.5. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Week 12 up to Week 24
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab Quarterly | Fremanezumab Monthly
Number analyzed (Participants) | 257 | 270 | 272
Participants | 3 | 1 | 3

16. Secondary Outcome: DB Period: Number of Participants With Potentially Clinically Significant Abnormal Urinalysis Laboratory Tests Results
Description: Criteria for potentially clinically significant abnormal urinalysis values included: urine glucose (milligrams/deciliter [mg/dL]): ≥2 unit increase from baseline, ketones (mg/dL): ≥2 unit increase from baseline, urine total protein (mg/dL): ≥2 unit increase from baseline, and haemoglobin ≥2 unit increase from baseline. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline up to Week 12
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab Quarterly | Fremanezumab Monthly
Number analyzed (Participants) | 277 | 276 | 285
Participants | 0 | 0 | 0

17. Secondary Outcome: OL Period: Number of Participants With Potentially Clinically Significant Abnormal Urinalysis Laboratory Tests Results
Description: Criteria for potentially clinically significant abnormal urinalysis values included: urine glucose (mg/dL): ≥2 unit increase from baseline, ketones (mg/dL): ≥2 unit increase from baseline, urine total protein (mg/dL): ≥2 unit increase from baseline, and haemoglobin ≥2 unit increase from baseline. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Week 12 up to Week 24
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab Quarterly | Fremanezumab Monthly
Number analyzed (Participants) | 262 | 271 | 274
Participants | 0 | 0 | 0

18. Secondary Outcome: DB Period: Number of Participants With Potentially Clinically Significant Abnormal Vital Signs Values
Description: Criteria for potentially clinically significant abnormal vital signs values included: pulse rate: ≤50 beats/minute (bpm) and decrease of ≥15 bpm, or ≥120 bpm and increase of ≥15 bpm; systolic blood pressure: ≤90 millimeters of mercury (mmHg) and decrease of ≥20 mmHg, or ≥180 mmHg and increase of ≥20 mmHg; diastolic blood pressure: ≤50 mmHg and decrease of ≥15 mmHg or ≥105 mmHg and increase of ≥15 mmHg; respiratory rate: <10 breaths/minute; and body temperature ≥38.3 degrees celsius and change of ≥1.1 degrees celsius. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline up to Week 12
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab Quarterly | Fremanezumab Monthly
Number analyzed (Participants) | 277 | 276 | 283
Participants | 9 | 8 | 8

19. Secondary Outcome: OL Period: Number of Participants With Potentially Clinically Significant Abnormal Vital Signs Values
Description: Criteria for potentially clinically significant abnormal vital signs values included: pulse rate: ≤50 bpm and decrease of ≥15 bpm, or ≥120 bpm and increase of ≥15 bpm; systolic blood pressure: ≤90 mmHg and decrease of ≥20 mmHg, or ≥180 mmHg and increase of ≥20 mmHg; diastolic blood pressure: ≤50 mmHg and decrease of ≥15 mmHg or ≥105 mmHg and increase of ≥15 mmHg; respiratory rate: <10 breaths/minute; and body temperature ≥38.3 degrees celsius and change of ≥1.1 degrees celsius. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Week 12 up to Week 24
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab Quarterly | Fremanezumab Monthly
Number analyzed (Participants) | 261 | 270 | 273
Participants | 10 | 14 | 8

20. Secondary Outcome: DB Period: Number of Participants With Shift From Baseline to Week 12 in Electrocardiogram (ECG) Parameters
Description: ECG parameters included: heart rate, PR interval, QRS interval, QT interval corrected using the Fridericia formula (QTcF), QT interval corrected using the Bazett's formula (QTcB) and RR interval. Shifts represented as Baseline - Week 12 value. Abnormal NCS indicated an abnormal but not clinically significant finding. Abnormal CS indicated an abnormal and clinically significant finding. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline, Week 12
Population: DB safety analysis set included all randomized participants who received at least 1 dose of study drug during the DB treatment period. Here, 'Overall number of participants analyzed' = participants with both baseline and Week 12 ECG findings.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab Quarterly | Fremanezumab Monthly
Number analyzed (Participants) | 258 | 271 | 270
Participants
  Normal - Normal | 199 | 218 | 212
  Normal - Abnormal NCS | 21 | 14 | 15
  Normal - Abnormal CS | 0 | 0 | 0
  Abnormal NCS - Normal | 10 | 19 | 12
  Abnormal NCS - Abnormal NCS | 28 | 20 | 31
  Abnormal NCS - Abnormal CS | 0 | 0 | 0
  Abnormal CS - Normal | 0 | 0 | 0
  Abnormal CS - Abnormal NCS | 0 | 0 | 0
  Abnormal CS - Abnormal CS | 0 | 0 | 0

21. Secondary Outcome: OL Period: Number of Participants With Shift From Baseline to Week 24 in ECG Parameters
Description: ECG parameters included: heart rate, PR interval, QRS interval, QT interval corrected using the Fridericia formula (QTcF), QT interval corrected using the Bazett's formula (QTcB) and RR interval. Shifts represented as Baseline - Week 24 value. Abnormal NCS indicated an abnormal but not clinically significant finding. Abnormal CS indicated an abnormal and clinically significant finding. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline, Week 24
Population: OL safety analysis set included all participants who received at least 1 dose of study drug during the OL treatment period. Here, 'Overall number of participants analyzed' = participants with both baseline and Week 24 ECG findings.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab Quarterly | Fremanezumab Monthly
Number analyzed (Participants) | 247 | 257 | 261
Participants
  Normal - Normal | 194 | 215 | 204
  Normal - Abnormal NCS | 15 | 5 | 15
  Normal - Abnormal CS | 0 | 0 | 1
  Abnormal NCS - Normal | 14 | 20 | 16
  Abnormal NCS - Abnormal NCS | 24 | 17 | 25
  Abnormal NCS - Abnormal CS | 0 | 0 | 0
  Abnormal CS - Normal | 0 | 0 | 0
  Abnormal CS - Abnormal NCS | 0 | 0 | 0
  Abnormal CS - Abnormal CS | 0 | 0 | 0

22. Secondary Outcome: DB Period: Number of Participants Who Received Concomitant Medications for Adverse Events
Description: Concomitant medications included: agents acting on the renin-angiotensin system, all other therapeutic products (for example: homeopathic preparation), allergens, analgesics, anesthetics, anti-parkinson drugs, antianemic preparations, antibacterials for systemic use, antibiotics and chemotherapeutics for dermatological use, antidiarrheals, intestinal antiinflammatory/antiinfective agents, antiemetic, antiepileptics, antifungals for dermatologiocal use, antigout preparations, antihemorrhagics, antihistamines for systemic use, antihypertensives, antiinflammatory and antirheumatic products, antimycotics for systemic use, antipruritics, antipsoriatics, antivirals for systemic use, beta blocking agents, blood substitutes and perfusion solutions, cardiac therapy, corticosteroids, cough and cold preparations, diagnostic radiopharmaceuticals, diuretics, thyroid therapy, urologicals, vaccines, psycoleptics, psycoanaleptics, ophthalmologicals, muscle relaxants, drugs used in diabetes etc.
Time Frame: Baseline up to Week 12
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab Quarterly | Fremanezumab Monthly
Number analyzed (Participants) | 277 | 276 | 285
Participants | 274 | 269 | 280

23. Secondary Outcome: OL Period: Number of Participants Who Received Concomitant Medications for Adverse Events
Description: as for outcome 22
Time Frame: Week 12 up to Week 24
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab Quarterly | Fremanezumab Monthly
Number analyzed (Participants) | 262 | 271 | 274
Participants | 262 | 266 | 270

ADVERSE EVENTS:
Time Frame: Baseline (Day 0) up to follow-up visit (Week 46)
Description: Safety analysis set included all participants who received at least 1 dose of study drug. AE data per system organ class (SOC) and preferred term (PT) were summarized collectively for both periods. 2 participants (1 with CM and 1 with EM) randomized to placebo but received Fremanezumab monthly dosing during double-blind treatment period. They were analyzed in the treatment arm per actual treatment received.
Arm/Group | Placebo | Fremanezumab Quarterly | Fremanezumab Monthly
All-Cause Mortality (participants affected / at risk) | 0/277 | 0/276 | 0/285
Serious Adverse Events (participants affected / at risk) | 13/277 | 10/276 | 11/285
Other Adverse Events (participants affected / at risk) | 88/277 | 90/276 | 81/285
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=277) | Fremanezumab Quarterly (N=276) | Fremanezumab Monthly (N=285)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Congenital diaphragmatic hernia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal tear (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Anal polyp (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Dengue fever (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Peritonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Respiratory fume inhalation disorder (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
International normalised ratio abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Angiomyxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/231 (1) | 0/229 (0) | 0/240 (0) — This is a gender-specific AE. Only female participants were at risk.
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/231 (1) | 0/229 (0) | 0/240 (0) — This is a gender-specific AE. Only female participants were at risk.
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Multiple sclerosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Optic neuritis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0/231 (0) | 1/229 (1) | 0/240 (0) — This is a gender-specific AE. Only female participants were at risk.
Endometriosis (Reproductive system and breast disorders) | 0/231 (0) | 0/229 (0) | 1/240 (1) — This is a gender-specific AE. Only female participants were at risk.
Menometrorrhagia (Reproductive system and breast disorders) | 0/231 (0) | 0/229 (0) | 1/240 (1) — This is a gender-specific AE. Only female participants were at risk.
Menorrhagia (Reproductive system and breast disorders) | 0/231 (0) | 1/229 (1) | 0/240 (0) — This is a gender-specific AE. Only female participants were at risk.
Metrorrhagia (Reproductive system and breast disorders) | 1/231 (1) | 0/229 (0) | 0/240 (0) — This is a gender-specific AE. Only female participants were at risk.
Vocal cord thickening (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=277) | Fremanezumab Quarterly (N=276) | Fremanezumab Monthly (N=285)
Injection site erythema (General disorders) | 24 (53) | 31 (66) | 32 (80)
Injection site induration (General disorders) | 16 (52) | 19 (41) | 18 (65)
Injection site pain (General disorders) | 10 (20) | 15 (42) | 14 (42)
Nasopharyngitis (Infections and infestations) | 32 (37) | 30 (41) | 25 (30)
Upper respiratory tract infection (Infections and infestations) | 10 (10) | 8 (11) | 16 (17)
Migraine (Nervous system disorders) | 21 (26) | 14 (15) | 12 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.

DOCUMENTS (2):
  • Study Protocol (2017-10-23): https://cdn.clinicaltrials.gov/large-docs/68/NCT03308968/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-13): https://cdn.clinicaltrials.gov/large-docs/68/NCT03308968/SAP_001.pdf